CLINICAL TRIAL: NCT00214916
Title: KULeuven Intensive Insulin Study in Pediatric Intensive Care Patients
Brief Title: Tight Glycemic Control With Intensive Insulin Therapy in PICU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Greet Van den Berghe (Other)
Responsible Party: Sponsor-Investigator, Greet Van den Berghe, Head of Dept and laboratory of Intensive Care Medicine, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PICU-insulin study; NCT00214916
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness
Keywords: Tight glycemic control with; intensive insulin treatment; versus conventional glycemic control; in infant or child in ICU
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): conventional insulin therapy (using Actrapid IV)
  Interventions: Drug: conventional insulin therapy (Actrapid IV only for excessive hyperglycemia)
- B (Experimental): intensive insulin therapy (using actrapid IV)
  Interventions: Drug: intensive insulin therapy (Actrapid IV to normoglycemia)

INTERVENTIONS:
Drug: intensive insulin therapy (Actrapid IV to normoglycemia) — intensive insulin therapy (Actrapid IV in continuous infusion to age-dependent normoglycemia)
  Other Names: Actrapid IV to normoglycemia
  Arms: B
Drug: conventional insulin therapy (Actrapid IV only for excessive hyperglycemia) — conventional insulin therapy (Actrapid IV in continuous infusion only to treat blood glucose levels exceeding 220 mg/dl)
  Other Names: Actrapid IV only for excessive hyperglycemia
  Arms: A

SUMMARY:
In a previous study, the investigators showed that tight blood glucose control with insulin during intensive care reduced morbidity and mortality in adult intensive care patients. Whether this intervention also improves prognosis of pediatric intensive care patients remains unknown. The current prospective, randomized, controlled study will asses the impact of intensive insulin therapy on outcome of patients in a pediatric intensive care unit. On admission patients will be randomly assigned to either strict normalization of blood glucose according age adjusted values or the conventional approach, in which insulin infusion is initiated only when blood glucose exceeds 215 mg/dl to maintain blood glucose levels between 180-200 mg/dl.

DETAILED DESCRIPTION:
Study type: Interventional study

Study design: single centre, prospective, randomized, active control, parallel assignment, efficacy study

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to the pediatric intensive care unit and anticipated to require intensive care for at least 24 hours

Exclusion Criteria:

* Expected stay < 24 hours
* Therapy restriction upon admission
* No informed consent
* Other study enrollment

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2004-10; Primary Completion 2008-02 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of inflammation | during ICU stay to day 5
duration of dependency on intensive care (days in ICU) | time in ICU

SECONDARY OUTCOMES:
Duration mechanical ventilation | during time in ICU
Organ failure/need for organ support | during time in ICU
mortality (safety endpoint) | during time in ICU
long-term follow-up study : focus on neurocognitive development (ethical approval granted) | 3 years (+/- 6 months) after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Greet Van den Berghe, MD,PhD, Study Director — Catholic University Leuven
Locations (1):
- Dep Intensive Care Medicine University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Derived] Verstraete S, Vanhorebeek I, Covaci A, Guiza F, Malarvannan G, Jorens PG, Van den Berghe G. Circulating phthalates during critical illness in children are associated with long-term attention deficit: a study of a development and a validation cohort. Intensive Care Med. 2016 Mar;42(3):379-392. doi: 10.1007/s00134-015-4159-5. Epub 2015 Dec 14. PMID 26667027
- [Derived] Sterken C, Lemiere J, Vanhorebeek I, Van den Berghe G, Mesotten D. Neurocognition after paediatric heart surgery: a systematic review and meta-analysis. Open Heart. 2015 Oct 29;2(1):e000255. doi: 10.1136/openhrt-2015-000255. eCollection 2015. PMID 26568832
- [Derived] Mesotten D, Gielen M, Sterken C, Claessens K, Hermans G, Vlasselaers D, Lemiere J, Lagae L, Gewillig M, Eyskens B, Vanhorebeek I, Wouters PJ, Van den Berghe G. Neurocognitive development of children 4 years after critical illness and treatment with tight glucose control: a randomized controlled trial. JAMA. 2012 Oct 24;308(16):1641-50. doi: 10.1001/jama.2012.12424. PMID 23101118
- [Derived] Gielen M, Mesotten D, Wouters PJ, Desmet L, Vlasselaers D, Vanhorebeek I, Langouche L, Van den Berghe G. Effect of tight glucose control with insulin on the thyroid axis of critically ill children and its relation with outcome. J Clin Endocrinol Metab. 2012 Oct;97(10):3569-76. doi: 10.1210/jc.2012-2240. Epub 2012 Aug 7. PMID 22872689
- [Derived] Gielen M, Mesotten D, Brugts M, Coopmans W, Van Herck E, Vanhorebeek I, Baxter R, Lamberts S, Janssen JA, Van den Berghe G. Effect of intensive insulin therapy on the somatotropic axis of critically ill children. J Clin Endocrinol Metab. 2011 Aug;96(8):2558-66. doi: 10.1210/jc.2010-3045. Epub 2011 Jun 1. PMID 21632816
- [Derived] Vlasselaers D, Mesotten D, Langouche L, Vanhorebeek I, van den Heuvel I, Milants I, Wouters P, Wouters P, Meyns B, Bjerre M, Hansen TK, Van den Berghe G. Tight glycemic control protects the myocardium and reduces inflammation in neonatal heart surgery. Ann Thorac Surg. 2010 Jul;90(1):22-9. doi: 10.1016/j.athoracsur.2010.03.093. PMID 20609741
- [Derived] Vlasselaers D, Milants I, Desmet L, Wouters PJ, Vanhorebeek I, van den Heuvel I, Mesotten D, Casaer MP, Meyfroidt G, Ingels C, Muller J, Van Cromphaut S, Schetz M, Van den Berghe G. Intensive insulin therapy for patients in paediatric intensive care: a prospective, randomised controlled study. Lancet. 2009 Feb 14;373(9663):547-56. doi: 10.1016/S0140-6736(09)60044-1. Epub 2009 Jan 26. PMID 19176240